CLINICAL TRIAL: NCT01108926
Title: Pharmacokinetics of Tenofovir and Tenofovir-diphosphate, Emtricitabine and Emtricitabine-triphosphate, and Efavirenz Once Daily Over 10 Days Following Drug Intake Cessation in Healthy Volunteers
Brief Title: PK of Tenofovir, Emtricitabine and Efavirenz in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Marta Boffito, St Stephen's AIDS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 035; 2009-018055-16 (EudraCT Number)
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infection; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Experimental): All Subjects will receive the same intervention
  Interventions: Drug: Atripla®

INTERVENTIONS:
Drug: Atripla® — All subjects will be administered Atripla® (tenofovir 245 mg plus emtricitabine 200 mg plus efavirenz 600 mg), one tablet orally once daily for 14 days
  Other Names: tenofovir = Viread®; emtricitabine = Emtriva® (formerly Coviracil); tenofovir + emtricitabine = Truvada®; efavirenz = Sustiva® and Stocrin®

SUMMARY:
The purpose of the study is to look at the levels of three HIV medications: tenofovir, emtricitabine, and efavirenz in blood after the drug intake has been stopped in order to understand how long these drugs persist in the blood. The study will specifically look at blood levels of these three drugs (taken as a 3-in-1 tablet) after taking them every day for 14 days.

This study is not randomised which means that all subjects will receive all study medications in the same order. You and the study doctor will know which study medications you are taking at all times during the study.

DETAILED DESCRIPTION:
The administration of combination antiretroviral therapy (cART) to HIV-infected patients has been associated with a dramatic reduction in AIDS-related morbidity and mortality [1-3].

The key to successful HIV drug treatment is adhering to the prescribed combination every day [2]. The approval of Atripla® (tenofovir/emtricitabine/efavirenz co-formulated in a single tablet) provides HIV care providers with a "one tablet once a day" therapy, making adherence much easier for patients.

However, in HIV therapy, successful adherence also means attention to intervals between doses or dietary restrictions. Ideally, to guarantee long-term virological response, HIV-infected patients should take their cART every day at the same time. However, cART is for life and doses can be forgotten or delayed.

Importantly, the 24-week 'Five-on-Two-off' (FOTO) study results were presented in November 2008; these showed that when HIV-infected patients stable (viral load < 50 copies/mL) on Atripla® were randomised to continue treatment daily or to stop taking it at weekends, no difference in maintenance of undetectable viral load was observed. Eighty percent in the control arm and 83% in the 'weekend off' arm had a viral load < 50 copies/mL [4]. This suggests that either the drugs' effects, or the drugs themselves, persist for a significant time following drug intake cessation. However, the persistence time and the inter-individual variability of this parameter for the components of Atripla® have not been clearly defined.

A drug's persistence in plasma or in cells depends on its half life. Long half-life antiretroviral agents may allow for missed or delayed doses, if concentrations are maintained at therapeutic levels until the next dose is taken. NRTI are pro-drugs and must be activated by different phosphorilation steps to be effective against HIV. Intracellular triphosphate (TP) metabolites have been shown to be characterized by long half lives. However, data on drug persistence are limited and whether drug doses can be omitted and dosing delayed is unknown.

Knowledge of the length of time the drug contained in the Atripla® formulation lasts would increase the confidence of doctors in this combination.

Importantly, triple regimen persistence should be investigated in order to provide information on the permissiveness (of forgotten or delayed doses) of the whole regimen rather than one single agent. Due to the simplicity of administering Atripla®, a study investigating the pharmacokinetic "forgiveness" of tenofovir and emtricitabine (in plasma and intracellularly) and plasma efavirenz would be readily performed in healthy volunteers and would provide information on how to advise HIV infected patients on delayed and missed doses.

Rationale for the pharmacogenomics analysis

Pharmacogenetics holds promise in HIV treatment because of the complexity and potential toxicity of multi antiretroviral drug therapies that are prescribed for long periods. Thus far, few candidate genes have been examined for a limited number of allelic variants, but a number of confirmed associations have already emerged.

From a public health perspective, as antiretroviral medications become increasingly available to racially and ethnically diverse populations worldwide, understanding the genetic structures of each population may allow us to anticipate the impact of adverse responses, even in groups that were not represented in drug registration trials.

The existing literature on pharmacogenetic determinants of antiretroviral drug exposure, drug toxicity, as well as genetic markers associated with the rate of disease progression underline the recent advances which occurred in the past few years.

However, it is expected that larger-scale comprehensive genome approaches will profoundly change the landscape of knowledge in the future. Additional studies are needed to assess the implications for long-term responses to antiretroviral agents.

For this reason we plan to collect a single blood sample from each participant in our intensive pharmacokinetic studies, such as this one, in order to be able to investigate the association between genetic polymorphisms in drug disposition genes (such as those encoding for cytochrome P450 isoenzymes or transmembrane transporters) and drug exposure. A candidate gene approach will be utilised to examine loci of interest. This procedure will provide potentially important information on genetic influences on plasma drug concentrations and give insight into how to improve the management of HIV-infected patients by individualising therapy. These studies will not be powered for genetic associations but will enable us to build a data base of genotype-phenotype. Prospective genetic studies would need to be planned based on these preliminary data.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 28 days prior to the baseline visit:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
5. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 12 weeks after the study
6. Willing to consent to their personal details being entered onto The Over volunteering Prevention Scheme (TOPS) database
7. Willing to provide photographic identification at each visit.
8. Registered with a GP in the UK

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Any significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B surface antigen and/or C antibodies
4. Positive blood screen for HIV-1 and/or 2 antibodies
5. Current or recent (within 3 months) gastrointestinal disease
6. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
7. Exposure to any investigational drug or placebo within 3 months of first dose of study drug
8. Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
9. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 12 weeks after the end of the treatment period
10. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of plasma tenofovir, emtricitabine and efavirenz | 24 days
  To assess the pharmacokinetics of plasma tenofovir and emtricitabine, and their active intracellular anabolites, tenofovir-diphosphate and emtricitabine-triphosphate, and plasma efavirenz over 10 days following drug intake cessation, in HIV negative healthy volunteers

SECONDARY OUTCOMES:
inter subject variability | 24 days
  To assess the inter subject variability in the concentrations of plasma tenofovir and emtricitabine, and their active intracellular anabolites, and plasma efavirenz following drug intake cessation
safety and tolerability of Atripla® | 24 days
  To assess the safety and tolerability of Atripla® over 14 days of administration in HIV negative healthy volunteers
pharmacogenetic | 24 days
  To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom

REFERENCES:
- See also: St Stephen's AIDS Trust website — http://www.ssat.org.uk/